CLINICAL TRIAL: NCT02034253
Title: Glutamate, Brain Connectivity and Duration of Untreated Psychosis
Acronym: DUP
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Dr. Adrianne C Lahti, Professor and Division Director of Behavioral Neurobiology, University of Alabama at Birmingham
Other Study IDs: 1R01MH102951 (NIH)
Record Dates: First submitted 2014-01-08; First posted 2014-01-13 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia; Psychosis; Schizoaffective Disorder
Keywords: duration of untreated psychosis; glutamate; functional connectivity; structural connectivity; schizophrenia; psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genes related to glutamate, n-acetyl-aspartate, dopamine, schizophrenia, and treatment response to antipsychotic medication will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- first episode psychosis: Unmedicated first episode psychosis patients that wish to enroll in a 16 week treatment regimen with the drug Risperidone.
  Interventions: Drug: Risperidone
- healthy demographic-matched controls: healthy controls will be matched to patients one to one based on: age, smoking status, parental socio-economic status, and gender. Healthy controls must be free from current or past Axis I mental disorders, 1st degree relative current or past Axis I mental disorders, and any other neurological conditions.

INTERVENTIONS:
Drug: Risperidone — Patients with psychosis will be provided a 16 week regimen of the antipsychotic drug Risperidone in accordance with standard care.
  Other Names: Risperdal
  Groups: first episode psychosis

SUMMARY:
The early stages of schizophrenia are associated with significant decreases in social and intellectual abilities, with more declines in chronic disease. Studies have identified relationships between duration of untreated psychosis (the duration between the onset of positive symptoms and treatment) and worse long term outcomes. However, the neurobiology of this phenomenon and its implications for response to antipsychotic medications remain poorly understood.

Glutamatergic excess altering brain connectivity might provide an explanation for why those with longer duration of untreated psychosis have worse clinical outcomes. The investigators propose to use neuroimaging to study 67 first episode psychosis subjects before and after sixteen weeks of treatment with risperidone, a common antipsychotic. We will measure (1) glutamate and (2) structural and functional brain connectivity and test the hypotheses that glutamatergic abnormalities are present in first episode patients and that longer duration of untreated psychosis is associated with greater connectivity abnormalities that set the stage for poor response to treatment. 67 demographic-matched controls will also be recruited as a comparison group - healthy controls will not receive antipsychotic medication.

The investigator's previous studies have made progress in the understanding of abnormalities in the glutamate system and brain connectivity in unmedicated patients with schizophrenia and modulation of these by antipsychotic medication. Two indices of glutamatergic dysfunction have been identified. While antipsychotic medications appear to modulate glutamate, the disturbance in the relationship between metabolites is not restored with treatment. In addition, the investigators found that both structural and functional connectivity abnormalities in unmedicated patients with schizophrenia predict patients' response to treatment.

To the investigator's knowledge, no other group has performed a study that uses a combination of complementary neuroimaging techniques that will allow generating a broad characterization of glutamatergic function and brain connectivity in first episode psychosis and change with treatment. The results of the proposed studies could suggest a mechanism by which the duration of untreated psychosis is associated with poor treatment response which might lead to new interventions to target the illness.

ELIGIBILITY:
Inclusion Criteria:

* Persons with first episode psychosis
* Healthy controls will be matched to first episode psychosis participants on a one to one basis

Exclusion Criteria:

* inability to understand and sign informed consent assessed by the Evaluation to sign Consent form
* diagnosable central nervous system illnesses
* poorly controlled acute or chronic medical conditions aside from psychosis
* history of head trauma with loss of consciousness for > 2 minutes
* active substance abuse or dependence (exclusive of nicotine dependence)
* suspected substance induced psychotic symptoms
* clinically significant symptoms of depression, hypomania, or mania
* patients concomitantly treated with drugs known to affect glutamate, such as: valproate, topiramate, gabapentin, levetiracetam, lamotrigine, lithium, and acamprosate

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The investigators expect to enroll a total of 67 male and female patients with first episode psychosis and 67 demographic matched controls.
  Among patients who participate in research at the University of Alabama at Birmingham (UAB) the approximate gender, ethnic and race distribution is 75% male and 25% female; 1% Hispanic and 99% Non-Hispanic; 54% White, 44% Black, and 1% Asian/Pacific Islander. The gender distribution is consistent with that observed in clinical populations with schizophrenia.
  Persons below the age of 17 and above the age of 35 are excluded to minimize the variance in cognitive functioning or brain connectivity that might be attributable to development rather than diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Comparison of indices of glutamate as measured by 1H-MRS in unmedicated first episode psychosis patients before and after antipsychotic treatment and with healthy controls. | Up to 5 years

SECONDARY OUTCOMES:
Comparison of structural and functional brain connectivity in first episode psychosis patients before and after antipsychotic treatment and healthy controls | Up to 5 years
  Structural brain connectivity (using diffusion tensor imaging) and functional brain connectivity (using resting state connectivity) will be compared between healthy controls and first episode psychosis patients. Additionally within first episode psychosis patients duration of untreated psychosis (DUP) will be correlated with both structural and functional brain connectivity to determine the impact of DUP on both metrics of brain connectivity.
Evaluation of the contribution of structural and functional connectivity to eventual antipsychotic treatment response in first episode psychosis patients. | Up to 5 years
  The investigators will evaluate the relationship between both structural brain connectivity (using diffusion tensor imaging) and functional brain connectivity (using resting state connectivity) before treatment and treatment response after 16 weeks of risperidone therapy in first episode psychosis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne C. Lahti, MD, Principal Investigator — University of Alabama at Birmingham, Department of Psychiatry
Locations (1):
- Sparks Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Maximo JO, Briend F, Armstrong WP, Kraguljac NV, Lahti AC. Higher-order functional brain networks and anterior cingulate glutamate + glutamine (Glx) in antipsychotic-naive first episode psychosis patients. Transl Psychiatry. 2024 Apr 10;14(1):183. doi: 10.1038/s41398-024-02854-7. PMID 38600117
- [Derived] Maximo JO, Briend F, Armstrong WP, Kraguljac NV, Lahti AC. Salience network glutamate and brain connectivity in medication-naive first episode patients - A multimodal magnetic resonance spectroscopy and resting state functional connectivity MRI study. Neuroimage Clin. 2021;32:102845. doi: 10.1016/j.nicl.2021.102845. Epub 2021 Sep 29. PMID 34662778
- [Derived] Maximo JO, Nelson EA, Armstrong WP, Kraguljac NV, Lahti AC. Duration of Untreated Psychosis Correlates With Brain Connectivity and Morphology in Medication-Naive Patients With First-Episode Psychosis. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Feb;5(2):231-238. doi: 10.1016/j.bpsc.2019.10.014. Epub 2019 Nov 9. PMID 31902581
- [Derived] Kraguljac NV, Anthony T, Skidmore FM, Marstrander J, Morgan CJ, Reid MA, White DM, Jindal RD, Melas Skefos NH, Lahti AC. Micro- and Macrostructural White Matter Integrity in Never-Treated and Currently Unmedicated Patients With Schizophrenia and Effects of Short-Term Antipsychotic Treatment. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 May;4(5):462-471. doi: 10.1016/j.bpsc.2019.01.002. Epub 2019 Jan 23. PMID 30852126
- [Derived] Sivaraman S, Kraguljac NV, White DM, Morgan CJ, Gonzales SS, Lahti AC. Neurometabolic abnormalities in the associative striatum in antipsychotic-naive first episode psychosis patients. Psychiatry Res Neuroimaging. 2018 Nov 30;281:101-106. doi: 10.1016/j.pscychresns.2018.06.003. Epub 2018 Jun 9. PMID 30286325